CLINICAL TRIAL: NCT06266741
Title: The Predictive Value of Lubricin in Patients With Infective Endocarditis
Status: Enrolling by invitation | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sevil Gulastı, Assistant Professor, Aydin Adnan Menderes University
Other Study IDs: NCT093509350936
Record Dates: First submitted 2023-10-25; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Infective Endocarditis
Keywords: Infective endocarditis; Lubricin; Glycoprotein; Procalcitonin
MeSH Terms: conditions — Endocarditis; Jacobs syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with infective endocarditis: Patients between the ages of 18-65 diagnosed with infective endocarditis according to the Duke criteria
  Interventions: Diagnostic Test: Lubricin
- Patients without infective endocarditis: Patients between the ages of 18-65 without diagnosed with infective endocarditis according to the Duke criteria
  Interventions: Diagnostic Test: Lubricin

INTERVENTIONS:
Diagnostic Test: Lubricin — Plasma lubricin levels can potentially serve as a biomarker in situations like endocardial injury and infection.

SUMMARY:
The main goal of this study is to evaluate the predictability of the disease by measuring the serum lubricin levels in patients with infective endocarditis and in non-patients

DETAILED DESCRIPTION:
Infective endocarditis is a challenging disease with a wide range of clinical presentations, making it difficult to diagnose. Diagnosis primarily relies on clinical suspicion based on symptoms. Blood cultures or other microbial tests confirming the presence of infection and echocardiography are supportive diagnostic tools. Another marker that may become valuable in the near future for diagnosing infective endocarditis is Lubricin. Lubricin, a glycoprotein expressed by the PRG4 gene, has been found to have significantly elevated levels in the plasma of animals with damaged or infected heart valves compared to healthy animals. Furthermore, plasma lubricin levels can potentially serve as a biomarker in situations like endocardial injury and infection. Lubricin and Procalcitonin will be studied from the blood samples routinely collected. During this academic study, procalcitonin and lubricin values will be measured by investigators. Thus, the sensitivity and specificity of the Lubricin parameter in patients with infective endocarditis will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be between 18 and 65 years old
* Patients diagnosed with infective endocarditis according to the Duke criteria

Exclusion Criteria:

- The patient being pregnant

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Along with 30 healthy individuals, 30 patients between the ages of 18 and 65 who meet the Duke criteria and do not receive antibiotic treatment due to infective endocarditis will be examined. Pregnant women will not be included in the study. During this examination, procalcitonin and lubricin values will be measured.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-11 (Estimated); Primary Completion 2024-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Valve damage indicative sign in infective endocarditis | through study completion, an average of 2 years
  Concentration of Lubricin parameter have a determinative role in patients with infective endocarditis

CONTACTS AND LOCATIONS:
Locations (1):
- Sevil Gulasti, Aydin, Zafer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the results of the statistical analysis of all collected data will be shared
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Delgado V, Ajmone Marsan N, de Waha S, Bonaros N, Brida M, Burri H, Caselli S, Doenst T, Ederhy S, Erba PA, Foldager D, Fosbol EL, Kovac J, Mestres CA, Miller OI, Miro JM, Pazdernik M, Pizzi MN, Quintana E, Rasmussen TB, Ristic AD, Rodes-Cabau J, Sionis A, Zuhlke LJ, Borger MA; ESC Scientific Document Group. 2023 ESC Guidelines for the management of endocarditis. Eur Heart J. 2023 Oct 14;44(39):3948-4042. doi: 10.1093/eurheartj/ehad193. No abstract available. PMID 37622656
- [Background] Rajani R, Klein JL. Infective endocarditis: A contemporary update. Clin Med (Lond). 2020 Jan;20(1):31-35. doi: 10.7861/clinmed.cme.20.1.1. PMID 31941729
- [Background] Holland TL, Baddour LM, Bayer AS, Hoen B, Miro JM, Fowler VG Jr. Infective endocarditis. Nat Rev Dis Primers. 2016 Sep 1;2:16059. doi: 10.1038/nrdp.2016.59. PMID 27582414
- [Background] Richendrfer H, Jay GD. Lubricin as a Therapeutic and Potential Biomarker in Sepsis. Crit Care Clin. 2020 Jan;36(1):55-67. doi: 10.1016/j.ccc.2019.08.005. Epub 2019 Oct 21. PMID 31733682
- [Background] Solakyildirim K, Li Y, Bayer AS, Sullam PM, Xiong YQ, Lebrilla CB, Bensing BA. Proteoglycan 4 (lubricin) is a highly sialylated glycoprotein associated with cardiac valve damage in animal models of infective endocarditis. Glycobiology. 2021 Dec 18;31(11):1582-1595. doi: 10.1093/glycob/cwab095. PMID 34459483